CLINICAL TRIAL: NCT00633685
Title: Predictors of Treatment Response to Fluoxetine in PTSD Following a Recent History of War Zone Stress Exposure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TEMPVA Research Group, Inc. (Other)
Collaborators: C.R.Darnall Army Medical Center (U.S. Federal Agency); Central Texas Veterans Health Care System (Other); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Paul B. Hicks, M.D., Ph.D./Associate Chief of Staff for Research, Central Texas Veterans Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR064845; PR064845
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-02

CONDITIONS: Posttraumatic Stress Disorder, Combat-related
Keywords: Posttraumatic Stress Disorder; Fluoxetine; Factors predicting response; Resilience; Pharmacologic augmentation strategies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Fluoxetine; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoxetine (Experimental): Receives Fluoxetine at 20-60 mg daily for 12 weeks in a flexible dosage schedule based upon clinical response
  Interventions: Drug: Fluoxetine; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Fluoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine will be administered at 20-60 mg daily for 12 weeks in a flexible dosage schedule based upon clinical response
  Other Names: Prozac
Drug: Placebo — Placebo will be empty gelatin capsules that are identical in size and shape to active treatment
  Other Names: Gelatin capsule

SUMMARY:
Three hundred (300) male or female outpatients, over 18 years of age, will be enrolled in this study to determine whether fluoxetine can be used as a treatment for Posttraumatic Stress Disorder in soldiers recently returning from combat exposure. There will be two phases to the study. In Phase I Fluoxetine + usual psychological care will be compared with Placebo + usual psychological care over a 12-week period. Subsequently, in Phase II all subjects will be offered the opportunity to enroll in a 20-week open-label trial on Fluoxetine. If response is inadequate, adjunctive treatment with either buspirone or bupropion will be offered. The investigational drugs are Fluoxetine, Buspirone and Bupropion. All are commercially available.

DETAILED DESCRIPTION:
While most soldiers exposed to the stresses of the war-zone exhibit psychological resilience, about one-fifth become psychological casualties of war. The fact that such a significant number of soldiers have difficulty adapting to life after war exposure suggests that we need to have well-defined treatments that are effective and cost-efficient. Currently, recommendations for first-line pharmacological management of Post-Traumatic Stress Disorder focus on the use of selective serotonin re-uptake inhibitors (SSRIs) such as fluoxetine. Despite this recommendation by the DoD/VA Clinical Practice Guidelines, there have not been any studies evaluating the effectiveness of these medications in patients that have recently been exposure to war-zone stressors. In fact, studies in Vietnam Era veterans have shown limited effectiveness of SSRIs for PTSD. In addition, there is very limited information available to understand the factors that influence whether a particular soldier will respond to treatment with an SSRI. This study is designed to determine whether fluoxetine is an effective treatment for PTSD and associated conditions in soldiers with recent war-zone exposure, as well as determine whether response to SSRIs is related to the severity of the trauma exposure and PTSD symptoms, psychological resilience, adequacy of social supports (family, extra-military and military), post-deployment stressors and life adversity, or the degree of any cognitive impairment.

After informed consent is given, fluoxetine (150 subjects) or placebo (150 subjects) will be administered for 12 weeks in doses from 20 mg daily up to 60 mg daily to active duty soldiers who are already receiving usual psychological care in the Resilience and Restoration Center of the Carl R. Darnall Army Medical Center at Ft. Hood. At the conclusion of this initial phase of the study, all participants will receive fluoxetine in doses up to 80 mg daily for an additional 20 weeks. All participants will be regularly monitored to determine changes in their PTSD symptoms. If a subject does not have at least a 50% improvement after being given 80 mg daily of fluoxetine for 4 weeks, then they will be randomly assigned to also receive either bupropion SR (150 mg daily) or buspirone (up to 40 mg daily) in an attempt to amplify the response to fluoxetine. Statistical analyses will be used to determine which factors provided the greatest influence on the response to these medication trials.

Each subject will be asked to receive a physical exam, give medical history information, and receive a diagnostic interview prior to participation in the study. After being randomly assigned to treatment, subjects will have interview or questionnaire assessments at weeks 2, 4, 6, 8, 12, 16, 20, 24, 28 and 32. Based solely on the degree of response as measured by the PTSD Checklist (a questionnaire that will be administered at each study visit), the dosage of study medication fluoxetine or placebo capsules will be adjusted by a pre-determined schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran of the OEF/OIF war campaigns with violence exposure sufficient to qualify for a diagnosis of PTSD
2. DSM-IV diagnosis of Post-Traumatic Stress Disorder as determined by the CAPS.
3. Entry Total CAPS score of at least 65
4. No exposure to psychotropic medications except for zolpidem for at least two weeks (five weeks for fluoxetine) prior to the baseline assessments.
5. If female, a negative beta-human chorionic gonadotropin pregnancy test and willing to use oral contraceptives

Exclusion Criteria:

1. History of intolerance to fluoxetine
2. History of lack of responsivity to a 60 mg daily dose of fluoxetine
3. Current or past history of Bipolar Disorder or Schizophrenia
4. Diagnosis of Major Depressive Disorder, Obsessive-Compulsive Disorder, or Other Anxiety Disorder, unless PTSD is the principal focus of treatment and the onset of PTSD preceded that of the concurrent disorders
5. Significant history of suicidal or homicidal behavior/ideation
6. Substance dependence in the past 6 months
7. Serious general medical condition that would risk the patient being able to complete the pharmacological trial with fluoxetine
8. Concomitant use of other antidepressants, antipsychotics or mood stabilizers
9. If female, pregnancy or unwilling to use oral contraceptives
10. Participation in another research drug trial within 30-days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | 12-Weeks

SECONDARY OUTCOMES:
PTSD Symptom Checklist | Every follow-up encounter (weeks 2-32)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Hicks, M.D., Ph.D., Principal Investigator — Central Texas Veterans Health Care System
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States